CLINICAL TRIAL: NCT00699803
Title: Study of T-PRED(TM) Compared to Pred Forte(R)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CL-PKT-0312081-P
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-Pred (Active Comparator): Tobramycin prednisolone acetate combination
  Interventions: Drug: T-PRED
- Pred Forte (Active Comparator): Prednisolone acetate
  Interventions: Drug: Pred Forte

INTERVENTIONS:
Drug: T-PRED — T-PRED sterile ophthalmic solution
  Arms: T-Pred
Drug: Pred Forte — Pred Forte sterile ophthalmic solution
  Arms: Pred Forte

SUMMARY:
Study of T-PRED(TM) compared to Pred Forte(R)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

Exclusion Criteria:

* No active or adverse disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- T-Pred: Tobramycin prednisolone acetate combination
  T-PRED: sterile ophthalmic solution
- Pred Forte: Prednisolone acetate
  Pred Forte: sterile ophthalmic solution
Period: Overall Study
Arm/Group | T-Pred | Pred Forte
Started | 32 | 32
Completed | 30 | 26
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-Pred | Pred Forte | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.0) | 65.7 (10.9) | 66.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Aqueous Humor Prednisolone Acetate Concentration
Time Frame: 4 hours
Population: Analysis Population was defined as all participants who received investigational product and on whom successful anterior chamber tap were performed at the designated time point
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pred Forte: Prednisolone acetate
  T-PRED: sterile ophthalmic solution
Arm/Group | T-Pred | Pred Forte
Number analyzed (Participants) | 30 | 26
ng/mL | 102.5 (5.6) | 127.5 (66.7)

ADVERSE EVENTS:
Time Frame: 4 hours
Groups:
- T-Pred: Tobramycin prednisolone acetate combination
  T-PRED: sterile ophthalmic solution at the first time point
  Pred Forte: sterile ophthalmic solution at the first time point
- Pred Forte: Prednisolone acetate
  T-PRED: sterile ophthalmic solution at the second time point
  Pred Forte: sterile ophthalmic solution at the second time point
Arm/Group | T-Pred | Pred Forte
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.